CLINICAL TRIAL: NCT06969989
Title: Effectiveness of Boswellia Sacra Extract Compared to Sodium Hypochlorite and Saline as Root Canal Irrigants in Pulpectomy of Necrotic Primary Molars: A Randomized Clinical Study
Brief Title: Herbal Irrigation in Necrotic Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doha Essam El Gohary, DR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: irrigation in primary molars
Record Dates: First submitted 2025-05-01; First posted 2025-05-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Herbal Irrigation in Necrotic Primary Molars
Keywords: herbal irrigation
MeSH Terms: interventions — Sodium Hypochlorite; Saline Solution

STUDY DESIGN:
Intervention Model Description: Frankincense is one of the herbal products that was traditionally used in folk medicine in many cultures due to its antibacterial, analgesic, and anti-inflammatory characteristics. In recent studies, practitioners have started using Frankincense as an intracanal irrigant in permanent teeth, comparing it with the gold standard sodium hypochlorite.
  Based on the current knowledge, no clinical trials in literature have been performed to compare the effectiveness of Boswellia Sacra water extract versus sodium hypochlorite as a root canal irrigant in pulpectomy of necrotic primary molars.
Who Masked: Participant, Outcomes Assessor
Masking Description: statisticians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 % water extract of Boswellia Sacra (Experimental): Canal shaping will be done using and rotary files then 10 mL of the tested irrigant( 10 % water extract of Boswellia Sacra) will be used for lubrication, flushing of debris and canal disinfection via a plastic disposable syringe with a 30-gauge side vented needle will be used 2mm short from the working length.
  Interventions: Other: 10 % water extract of Boswellia Sacra
- 1 % Sodium Hypochlorite (Active Comparator): Canal shaping will be done using rotary files and 10 mL of the tested irrigant ( 1% NAOCL) will be used for lubrication, flushing of debris and canal disinfection via a plastic disposable syringe with a 30-gauge side vented needle will be used 2mm short from the working length.
  Interventions: Other: 1 % Sodium Hypochlorite
- 0.9 % saline (Placebo Comparator): Canal shaping will be done using rotary files and 10 mL of the tested irrigant ( 0.9 % saline)will be used for lubrication, flushing of debris and canal disinfection via a plastic disposable syringe with a 30-gauge side vented needle will be used 2mmshort from the working length.
  Interventions: Other: 0.9 % Normal Saline

INTERVENTIONS:
Other: 10 % water extract of Boswellia Sacra — Canal shaping will be done using and rotary files with aid of 10 mL of the tested irrigant( 10 % water extract of Boswellia sacra) for lubrication, flushing of debris and canal disinfection via a plastic disposable syringe with a 30-gauge side vented needle will be used 2mm short from the working length
  Arms: 10 % water extract of Boswellia Sacra
Other: 1 % Sodium Hypochlorite — Canal shaping will be done using and rotary files with aid of 10 mL of the tested irrigant ( 1 % NaOCl ) for lubrication, flushing of debris and canal disinfection via a plastic disposable syringe with a 30-gauge side vented needle will be used 2mm short from the working length
  Arms: 1 % Sodium Hypochlorite
Other: 0.9 % Normal Saline — Canal shaping will be done using and rotary files with aid of 10 mL of the tested irrigant (0.9 % saline) for lubrication, flushing of debris and canal disinfection via a plastic disposable syringe with a 30-gauge side vented needle will be used 2mm short from the working length
  Arms: 0.9 % saline

SUMMARY:
Frankincense is one of the herbal products that was traditionally used in folk medicine in many cultures due to its antibacterial, analgesic, and anti-inflammatory characteristics .In recent studies, practitioners have started using Frankincense as an intracanal irrigant in permanent teeth, comparing it with the gold standard sodium hypochlorite. Based on the current knowledge, no clinical trials in literature have been performed to compare the effectiveness of Boswellia Sacra water extract versus sodium hypochlorite as a root canal irrigant in pulpectomy of necrotic primary molars.

DETAILED DESCRIPTION:
Maintaining a healthy primary dentition is necessary for the proper development of the successors. Dental caries with pulpal involvement is one of the most widespread communicable diseases in children. Thus, in some instances, a pulpectomy procedure is essential to save the deciduous tooth from early extraction. As a result of the complex anatomy of root morphology and wide, apical foramen, a safe, potent irrigant is necessary to help disinfect the root canal system without harming the periapical tissues and the permanent tooth bud. Pulpectomy of primary teeth is indicated when the pulp tissue is irreversibly infected or necrotic due to caries or trauma. The treatment consists of extirpation of the pulp tissue, removal of organic debris with filing, and obturation of the canals with a suitable material .

The cleaning and shaping of the root canal process depends on a chemo-mechanical disinfection procedure, mechanically through canal shaping aiming to remove inflamed & necrotic pulps tissues and infected debris from the root canal system, and chemically by the use of chemical antibacterial irrigants to disinfect the root canals and cause an aggressive decrease in the bacterial load inside the root canal system . Effective irrigant delivery is a prerequisite to root canal disinfection and debris removal to Improve endodontic treatment outcomes. Several irrigation agents have been developed in response to chemical disinfection. However, sodium hypochlorite (NaOCl) remains the irrigant of choice due to its antibacterial nature, dissolving both necrotic and organic matter within the smear layer.

Preventing post-endodontic pain is essential for both patients and clinicians. Postoperative pain is common after root canal treatment. It is mainly attributed to mechanical, chemical, and microbiological factors, especially in teeth with nonvital pulps, usually occurring due to the extrusion of infected debris and fluids.

Microorganisms and their metabolites are intimately related to the etiology of pulp and periapical pathology. The removal/elimination of pulp remnants, microorganisms, and byproducts is important for endodontic treatment success. Lipopolysaccharide (LPS), generally referred to as endotoxin, is present in the outer cell membranes of Gram-negative bacteria and is released during cell division or cell death, being one of the most important virulence factors involved in the development and maintenance of periapical inflammation and clinical symptomatology. Special attention has been given to the complete removal/neutralization of endotoxin from infected root canals The direction towards the usage of herbal products has gained great attention in recent years. The advantages they offer make them regarded as promising substitutions for synthetic chemical agents. Different essential oils with various purposes have been discovered and used for about 43 species of Boswellia. Boswellia sacra, one of the frankincense family, has been recommended to cure wounds, sores, and ulcers. In addition. Frankincense water extract has been utilized by ArabAfrican and Middle Eastern nations to alleviate cough, sore throat, and different gastrointestinal problems.

The Omani Luban, Oleo-Gum Resin of Boswellia sacra Flueck have been tested via in vitro studies showing antibacterial efficiency for its essential oils. Another research declared its promising chelating property in comparison to 17 % EDTA when used as an intracanal irrigant. Furthermore, another study revealed the regenerating power of boswellic acids for bone healing after endodontic surgeries.

ELIGIBILITY:
Inclusion Criteria:

Mandibular primary molars with deep caries and necrotic pulp.

* Mobility independent from normal physiological exfoliation
* Pain on percussion.
* Presence of fistula or furcation abscess.
* Restorable tooth
* Radiolucency in periapical or furcation area.
* Widening of PDL space or loss of lamina dura continuity.
* At least 2/3 root is present

Exclusion Criteria:

* Uncooperative children to avoid time waste and attrition bias.
* Children with systemic disease as some systemic diseases may affect the outcome.
* Lack of informed consent by the child patient's parent to be approved ethically.
* Refusal of participation.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | Records will be taken before the procedure then ( 6/ 12/ 24 hours) post procedure completion
  Visual Analog Pain Rating Scale will be explained to the children, and preoperative pain scores will be recorded. After completion post operative pain scores will be recorded as follows ( 6 / 12 / 24 hours )after the procedure.
  Visual Analog Pain Rating Scale with scores Categorical(0-10) - 0 no pain - 1-3 mild pain - 4-6 moderate pain - 7-10 severe pain.

SECONDARY OUTCOMES:
Bacterial count measure | S1 sample will be taken before chemo-mechanical preparation post access cavity . s2 samplewill be taken during the procedure immediately post completion of chemo-mechanical preparation
  Microbiological analysis by aerobic and anaerobic bacterial culture. A Pre-preparation sample (S1) will be taken from the root canal just after the tooth is accessed. Three sterile paper points (size 15) will be introduced in the largest canal 1mm shorter than the working length predetermined by the apex locator. The paper points will be left in the canal for at least one minute, then transferred to a sterile Eppendorf tube containing the transfer media Brain heart infusion (BHI) broth, placed in an ice box and transferred for culture.
  Post-instrumentation samples (s2) will be taken with three sterile paper points (size 15) introduced in the largest canal 1mm shorter than the working length which predetermined by the apex locator. The paper points will be left in the canal for for at least one minute, then transferred to a sterile Eppendorf tube containing the transfer media Brain heart (BHI) broth, placed in an ice box and transferred for culture.
Amount of endotoxins | S1 sample will be taken before chemo-mechanical preparation after access cavity is done . s2 sample will be taken during the procedure immediately post the completion of chemo-mechanical preparation.
  The three sterile paper points (size 15) will be introduced in the largest canal 1mm shorter than the working length predetermined by the apex locator. The paper points will be left in the canal for at least one minute then placed in a sterile empty Eppendorf tube for further Enzyme-linked immunosorbent assay (ELISA) to determine the number of endotoxins.
  Post-instrumentation samples (s2) will be taken as previously described for (s1).Three sterile paper points (size 15) will be introduced in the largest canal 1mm shorter than the working length predetermined by the apex locator. The paper points will be left in the canal for at least one minute then placed in a sterile empty Eppendorf tube for further Enzyme-linked immunosorbent assay (ELISA) to determine the number of endotoxins.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Dentistry and Dental Public Health Department - Faculty of Dentistry, Cairo University - Egypt., Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD might be shared on reasonable request